CLINICAL TRIAL: NCT00665587
Title: Surgical Treatment of Atrial Fibrillation - Prospective Randomized Study
Brief Title: AMAZING PRAGUE (PRAGUE-12)
Acronym: AmP
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Prof. MUDr. Zbynek Straka, CSc., Kralovske Vinohrady University Hospital
Other Study IDs: 121402
Record Dates: First submitted 2008-04-23; First posted 2008-04-24 (Estimated); Last update posted 2008-04-24 (Estimated); Status verified 2008-04

CONDITIONS: Atrial Fibrillation; Restore of Sinus Rhythm; Post-Operative Complications
Keywords: Atrial fibrillation; Maze procedure; Mid-term results; Long-term results; Surgical ablation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Maze Procedure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- A = MAZE: Patients indicated to a cardiac surgery (bypass, valve repair or combinated surgery)with documented atrial fibrillation in 6 preoperative months undergo the operation together with MAZE procedure
  Interventions: Procedure: Cox-MAZE III
- B = non-MAZE: Patients indicated to a cardiac surgery (bypass, valve repair or combinated surgery)with documented atrial fibrillation in 6 preoperative months undergo the operation (without MAZE procedure).

INTERVENTIONS:
Procedure: Cox-MAZE III — Maze procedure according to standards of the department
  Groups: A = MAZE

SUMMARY:
Aim of the project is to assess the long-time clinical impact of surgical ablation (MAZE procedure) on patients who suffer from atrial fibrillation but are indicated to a cardiac surgery for other predominant cardiac diagnosis (heart valve surgery, coronary revascularization or combined surgery). In recent years, those patients are more and more frequently indicated to some type of MAZE procedure, without the real benefit of this procedure for patients has been assessed with an enough large, randomized study. Even though it is well known, that MAZE procedures declines the early postoperative incidence of atrial fibrillation, convincing data about its mid-term and long-term impact on patients and about the appearance of recidives of atrial fibrillation in long-time horizon are still missing. Our hypothesis assumes, that MAZE procedure will significantly decrease the appearance of atrial fibrillation one year after the operation, without increasing mortality or incidence of serious postoperative complications in thirty postoperative days.

ELIGIBILITY:
Inclusion Criteria:

* indication to a cardiac surgery (coronary bypass, valve repair, others or combination of those)
* atrial fibrillation (paroxysmal, persistent or permanent) present or documented in last 6 month before the operation
* signed informed consent

Exclusion Criteria:

* rejection of signing the informed consent with randomization
* emergent surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who suffer from atrial fibrillation (documented AF in 6 month before the surgery) but are indicated to a cardiac surgery for other predominant cardiac diagnosis (heart valve surgery, coronary revascularization or combined surgery)
Sampling Method: Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2007-06; Primary Completion 2009-06 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
presence of sinus rhythm | 1 year after surgery
death, myocardial infarction, vascular cerebral attack, renal failure with a need of haemodyalisis | 30 postoperative days

SECONDARY OUTCOMES:
mortality, presence of sinus rhythm, serious complications- bleeding, vascular cerebral attack, heart failure, anticoagulation, anti-arrhytmics, pacemaker or ICD implantation, catether ablation... | 1,3,5 months 1,5 years after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Zbynek Straka, Prof.,MUDr.,CSc., Principal Investigator — Charles University, Prague
Locations (3):
- Czechia (3):
  - Cardiosurgery Department of University Hospital in Pilsen, Pilsen
  - Cardiocentre of Kralovske Vinohrady University Hospital, Prague
  - Cardiology department of Masarykova Hospital Usti nad Labem, Ústí nad Labem